CLINICAL TRIAL: NCT02447913
Title: To Observe the Effectiveness of a Demand-Side Financing Project in Increasing Demand and Utilization of Contraceptives for Birth Spacing Among Women From Poorest Two Quintiles in Faisalabad District of Pakistan
Brief Title: Integrating Family Planning With Immunization to Improve Maternal and Child Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Greenstar Social Maketing (Industry)
Collaborators: David and Lucile Packard Foundation (Other); Population Services International (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Grant #2011-37081
Record Dates: First submitted 2015-05-05; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Contraception
Keywords: Family planning; Voucher; Immunisations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voucher (Experimental)
  Interventions: Behavioral: Voucher
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Voucher — Introduction of vouchers will improve uptake of family method as well as child immunization.
  Incentivizing the providers to improve their counseling skills will improve the provider client relationship and better compliance of Family planning method
  Arms: Voucher

SUMMARY:
The proposed project will help in assessing the effectiveness of a demand-side financing project that provides family planning services bundled in a package of postnatal care and infant immunization services. This approach will use postnatal and infant health as a gateway to family planning - building confidence among the client and her influencers in the provider and repositioning family planning as part of a continuum of care to ensure the health of the mother and the infant. Vouchers will help in creating demand among poor women for the Family planning and child immunization. Also incentivizing providers against each voucher will help in improving their counselling skills as they will spend more time with voucher clients resulting is a satisfied client and better compliance with Family planning methods.

DETAILED DESCRIPTION:
Study hypothesis: Contraceptive Prevalence Rate will increase up to 20% from the baseline to end line survey in the intervention area .Contraceptive Prevalence Rate will increase by 5% between baseline and end line survey in the control area.

Ethics approval: The study has been approved by Population Services International Research Ethics Board.

Study design: This is a quasi experimental design. The study is a single center.

Primary study design: Interventional Trial setting: Community. Interventions: Introduction of vouchers will improve uptake of family method as well as child immunization.

Incentivizing the providers to improve their counseling skills will improve the provider client relationship and better compliance of Family planning method.

Intervention Type: Behavioral Primary outcome measures: Number of women who took up modern, reversible contraceptive methods ,number of women who availed postnatal care and number of women whose infants were immunized among the two poorest quintiles.

Secondary outcome measures: Improve the quality of family planning service provision in private sector health facilities serving low-income women.

Eligibility

Participant inclusion criteria - Participant type: Other. Participant inclusion criteria - Description: Women who are married in their reproductive age group i-e 15 to 49 years and who have given birth to a child within past one month.

Participant inclusion criteria - Target number of participants: 28000. Participant exclusion criteria: Women who are not married and are not in their reproductive age group i-e 15-49 years and who has not given birth within past 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Women who are married in their reproductive age group i-e 15 to 19 years and who have given birth to a child within past one month

Exclusion Criteria:

* Women who are not married and are not in their reproductive age group i-e 15-49 years and who has not given birth within past 1 month

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28000 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
number of women who used modern,reversible contraceptive methods | 2-3 years
number of women who had postnatal care | 2-3 years
number of women whose infants had immunizations | 2-3years

SECONDARY OUTCOMES:
Improve the quality of family planning service provision in private sector health facilities as judged by client satisfaction criteria | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Memon, Principal Investigator — Greenstar Social Marketing
Locations (1):
- Faisalabad, Punjab Province, Pakistan